CLINICAL TRIAL: NCT00473590
Title: A Randomized, Blinded, Placebo-Controlled, Multicenter, Phase II Study of Bevacizumab in Combination With Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Bevacizumab in Combination With Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma (AMBER)
Acronym: AMBER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVF4064g
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: Avastin; AMBER; Myeloma; Velcade
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bevacizumab; Bortezomib

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Bortezomib + bevacizumab (Experimental): Participants received bortezomib 1.3 mg/m^2 administered as a 3- to 5-second bolus intravenous injection on Days 1, 4, 8, and 11 of a 21-day cycle for a maximum of eight cycles and bevacizumab 15 mg/kg administered by intravenous infusion on the first day of each 21-day cycle during the blinded treatment phase. After completion of 8 cycles, participants could continue to receive bevacizumab as monotherapy until disease progression.
  Interventions: Drug: Bevacizumab; Drug: Bortezomib
- Bortezomib + placebo (Active Comparator): Participants received bortezomib 1.3 mg/m^2 administered as a 3- to 5-second bolus intravenous injection on Days 1, 4, 8, and 11 of a 21-day cycle for a maximum of eight cycles and placebo intravenous infusion on the first day of each 21-day cycle during the blinded treatment phase. At the completion of the 8-cycle treatment phase, participants entered the observation phase until disease progression.
  Interventions: Drug: Bortezomib; Drug: placebo

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg administered by intravenous infusion
  Arms: Bortezomib + bevacizumab
Drug: Bortezomib — 1.3 mg/m^2 administered by intravenous bolus injection
Drug: placebo — Intravenous repeating dose
  Arms: Bortezomib + placebo

SUMMARY:
This is a randomized, blinded, placebo-controlled, multicenter, Phase II study designed to provide a preliminary assessment of the safety and efficacy of combining bevacizumab with bortezomib in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Previously diagnosed with multiple myeloma
* Relapsed or refractory multiple myeloma with disease progression following one to three prior treatment regimens
* Measurable multiple myeloma disease

Exclusion Criteria:

* Grade ≥ 2 peripheral neuropathy
* Use of corticosteroids within 21 days prior to Day 1
* Use of other anti-myeloma therapy within 21 days prior to Day 1
* Intolerance to bortezomib or compounds containing boron
* Life expectancy of < 12 weeks
* Current, recent, or planned participation in an experimental drug study
* Active malignancy other than multiple myeloma within 5 years before screening
* Prior treatment with bevacizumab
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF)
* Decreased left ventricular function at study entry
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Significant vascular disease or recent peripheral arterial thrombosis within 6 months prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, including placement of a vascular access device within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture (for pathologic bone fractures consistent with multiple myeloma, patients may be eligible if no treatment is planned)
* Albuminuria
* Known hypersensitivity to any component of bevacizumab
* Pregnancy (positive pregnancy test) or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia (Ginny) Paton, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase II, randomized, blinded, placebo-controlled, multicenter study designed to provide a preliminary assessment of the safety and efficacy of combining bevacizumab with bortezomib in patients with relapsed or refractory multiple myeloma starting 11 July 2007 and completing 9 November 2009.
Groups:
- BORT + P: Participants received bortezomib 1.3 mg/m^2 administered as a 3- to 5-second bolus intravenous injection on Days 1, 4, 8, and 11 of a 21-day cycle for a maximum of eight cycles and placebo intravenous infusion on the first day of each 21-day cycle during the blinded treatment phase. At the completion of the 8-cycle treatment phase, participants entered the observation phase until disease progression.
- BORT + BV: Participants received bortezomib 1.3 mg/m^2 administered as a 3- to 5-second bolus intravenous injection on Days 1, 4, 8, and 11 of a 21-day cycle for a maximum of eight cycles and bevacizumab 15 mg/kg administered by intravenous infusion on the first day of each 21-day cycle during the blinded treatment phase. After completion of 8 cycles, participants could continue to receive bevacizumab as monotherapy until disease progression.
Period: Overall Study
Arm/Group | BORT + P | BORT + BV
Started | 53 | 49
Treated | 52 | 48
Safety Population | 50 (2 patients received at least 1 bevacizumab dose & were analyzed as bevacizumab-treated patients) | 50
Completed | 8 (Continuing on study as of the data cutoff date of 9 November 2009.) | 11 (Continuing on study as of the data cutoff date of 9 November 2009.)
Not Completed | 45 | 38
Not completed — Adverse Event | 3 | 3
Not completed — Death | 4 | 2
Not completed — Progression not resulting in death | 24 | 20
Not completed — Non-protocol-specified therapy | 7 | 5
Not completed — Physician Decision | 2 | 4
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BORT + P | BORT + BV | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.2) | 65.6 (9.3) | 65.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 30 | 29 | 59

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With an Overall Response
Description: Overall response was defined as a stringent complete response, complete response, very good partial response, or partial response (sCR, CR, VGPR, and PR, respectively) determined on two consecutive assessments ≤ 6 weeks apart and before the initiation of any new anti-tumor therapy, as assessed by the investigator using the International Myeloma Working Group's (IMWG's) uniform response criteria. Patients without a post-baseline response assessment or who died prior to their first scheduled response assessment were considered non-responders.
Time Frame: From randomization to the end of study (clinical cut-off; up to 116 weeks).
Population: Randomized Patients
Measure: Number; unit: participants
Arm/Group | BORT + P | BORT + BV
Number analyzed (Participants) | 53 | 49
participants | 23 | 25

2. Secondary Outcome: Percentage of Participants With an Overall Response
Description: Overall response was defined as a stringent complete response, complete response, very good partial response, or partial response (sCR, CR, VGPR, and PR) determined on two consecutive assessments ≤ 6 weeks apart and before the initiation of any new anti-tumor therapy, as assessed by the investigator using the IMWG's uniform response criteria. Patients without a post-baseline response assessment or who died prior to their first scheduled response assessment were considered non-responders.
Time Frame: From randomization to the end of study (clinical cut-off; up to 116 weeks).
Population: Randomized Patients
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BORT + P | BORT + BV
Number analyzed (Participants) | 53 | 49
Percentage of Participants | 43.4 [30.1 to 57.7] | 51.0 [36.3 to 65.2]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the initial response to disease progression or death on study. Disease progression was determined by the investigator using the IMWG's uniform response criteria and defined as an increase of ≥25% from best response in: Serum M-protein and/or Urine M-protein and/or Marrow plasma cells; or new or increased plasmacytomas or bone lesions; or hypercalcemia due to myeloma. Duration of response was estimated using Kaplan-Meier. For patients who had not progressed or died, duration of response was censored at the date of the last response assessment.
Time Frame: From randomization to the end of study (clinical cut-off; up to 116 weeks).
Population: Randomized Patients with an overall response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BORT + P | BORT + BV
Number analyzed (Participants) | 23 | 25
Months | 6.0 [4.86 to 8.31] | 6.9 [4.73 to 11.83]
Statistical Analysis 1: Comparison: BORT + P vs BORT + BV; Stratified analysis; Test type: Superiority or Other; p = 0.9179, Log Rank; The strata were number of prior cancer treatments (1, > 1) and β2-microglobulin level (< 3.5, ≥ 3.5 mg/L); Hazard Ratio (HR) = 0.956, 95% CI 2-sided [0.404 to 2.261] — The hazard ratios were estimated using Cox regression
Statistical Analysis 2: Comparison: BORT + P vs BORT + BV; Unstratified analysis; Test type: Superiority or Other; p = 0.6665, Log Rank — The tests were exploratory because patients were not randomized to the two arms with respect to response status; Hazard Ratio (HR) = 0.836, 95% CI 2-sided [0.369 to 1.893] — The hazard ratios were estimated using Cox regression

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the duration of time from randomization until death from any cause. All deaths were included, whether they occurred on study treatment or following treatment discontinuation. Overall survival was estimated using Kaplan-Meier. For patients who had not died, overall survival was censored at the date that the patient was last known to be alive.
Time Frame: From randomization until death from any cause, up until the end of study (clinical cut-off; up to 116 weeks).
Population: Randomized Patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BORT + P | BORT + BV
Number analyzed (Participants) | 53 | 49
Months | 24.0 [15.24 to NA] — Upper limit of 95% CI not estimable due to too few events at the time of analysis. | NA [NA to NA] — The median duration of overall survival in the BORT + BV arm was not estimable, as too few events had been observed
Statistical Analysis 1: Comparison: BORT + P vs BORT + BV; Stratified analysis; Test type: Superiority or Other; p = 0.3134, Log Rank; Hazard Ratio (HR) = 0.633, 95% CI 2-sided [0.258 to 1.552] — The hazard ratios were estimated using Cox regression. The strata were number of prior cancer treatments (1, > 1) and β2-microglobulin level (< 3.5, ≥ 3.5 mg/L)
Statistical Analysis 2: Comparison: BORT + P vs BORT + BV; Unstratified analysis; Test type: Superiority or Other; p = 0.2634, Log Rank; Hazard Ratio (HR) = 0.608, 95% CI 2-sided [0.251 to 1.468] — The hazard ratios were estimated using Cox regression

5. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from randomization to disease progression or death on study from any cause within 30 days of the last response assessment. Disease progression was determined by the investigator using the International Myeloma Working Group's (IMWG) uniform response criteria. Median PFS was estimated using Kaplan-Meier methodology. For patients who were alive at the time of the analysis and whose disease had not yet progressed, PFS was censored at the time of the last response assessment.
Time Frame: From randomization to disease progression or death on study (up to 116 weeks).
Population: Randomized Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BORT + P | BORT + BV
Number analyzed (Participants) | 53 | 49
months | 5.1 [4.17 to 7.20] | 6.2 [4.40 to 8.54]
Statistical Analysis 1: Comparison: BORT + P vs BORT + BV; The null hypothesis was that there was no difference between the 2 treatment groups. The alternative hypothesis was that progression-free survival was longer in the BORT + BV group. Stratified Analysis; Test type: Superiority or Other; p = 0.2804, Log Rank; The analysis was stratified for number of prior cancer treatments (1, > 1) and β2-microglobulin level (< 3.5, ≥ 3.5 mg/L); Hazard Ratio (HR) = 0.743, 95% CI 2-sided [0.432 to 1.276] — The hazard ratio was estimated using Cox regression. The hazard ratio is relative to BORT + P
Statistical Analysis 2: Comparison: BORT + P vs BORT + BV; Unstratified Analysis; Test type: Superiority or Other; p = 0.2009, Log Rank; Hazard Ratio (HR) = 0.713, 95% CI 2-sided [0.424 to 1.200] — Hazard ratio relative to BORT + P was estimated using Cox regression

6. Secondary Outcome: Number of Participants With Selected Adverse Events (AEs)
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0. All serious adverse events are listed in the Adverse Event Reporting section.
Time Frame: Participants were monitored for AEs from initiation of treatment to 30 days after treatment termination (up to 122 weeks).
Population: Safety population: all patients who were randomized and received any amount of study treatment. Two patients who randomized to the BORT + P arm received at least 1 dose of bevacizumab and were analyzed as bevacizumab-treated patients. Therefore, the safety analysis included 50 patients in the BORT + P arm and 50 patients in the BORT + BV arm.
Measure: Number; unit: Participants
Arm/Group | BORT + P | BORT + BV
Number analyzed (Participants) | 50 | 50
Participants
  Arterial thromboembolic events (any grade) | 0 | 1
  Bleeding other than pulmonary or CNS (Grade >=3) | 1 | 2
  Febrile neutropenia (any grade) | 1 | 1
  Gastrointestinal Perforation (Any Grade) | 1 | 0
  Hypertension (Grade >= 3) | 0 | 8
  Left Ventricular Systolic Dysfunction (Grade >= 3) | 1 | 0
  Neutropenia (Grade >= 3) | 6 | 10
  Osteonecrosis of the Jaw | 0 | 1
  Peripheral Neuropathy (Grade >= 3) | 7 | 8
  Pulmonary and CNS Bleeding (Any Grade) | 0 | 1
  Thrombocytopenia (Grade >= 3) | 15 | 15
  Vernous Thromboembolic Events (Grade >=3) | 1 | 0

ADVERSE EVENTS:
Time Frame: Participants were monitored for AEs from initiation of treatment to 30 days after treatment termination.
Description: Two patients who were randomized to the BORT + P arm received at least one dose of bevacizumab during the study and were analyzed as bevacizumab-treated patients. Therefore, 50 patients in the BORT + P arm and 50 patients were included in the BORT + BV arm in the safety analysis.
Arm/Group | BORT + P | BORT + BV
Serious Adverse Events (participants affected / at risk) | 26/50 | 24/50
Other Adverse Events (participants affected / at risk) | 41/50 | 43/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BORT + P (N=50) | BORT + BV (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Atrial Flutter (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Vertigo (Cardiac disorders) | 0 | 1
Ulcerative Keratitis (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal Perforation (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Drug Withdrawal Syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Abscess Jaw (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial Infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Ureteritis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 3 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BORT + P (N=50) | BORT + BV (N=50)
Anaemia (Blood and lymphatic system disorders) | 6 | 9
Neutropenia (Blood and lymphatic system disorders) | 6 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 14
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Fatigue (General disorders) | 3 | 6
Neuralgia (Nervous system disorders) | 6 | 10
Neuropathy Peripheral (Nervous system disorders) | 8 | 8
Hypertension (Vascular disorders) | 2 | 10
Pyrexia (General disorders) | 3 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 6
Urinary Tract Infection (Infections and infestations) | 3 | 2
Headache (Nervous system disorders) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.